CLINICAL TRIAL: NCT04552990
Title: Jet-Injection Assisted Photodynamic Therapy for Basal Cell Carcinoma
Brief Title: Use of Jet-injection in Photodynamic Therapy for Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-270
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: BCC; BCC - Basal Cell Carcinoma; Basal Cell Carcinoma; Basal Cell Cancer; Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma
Keywords: Superficial BBC; Nodular BBC; Superficial Basal Cell Carcinoma; Nodular Basal Cell Carcinoma; BCC; Basal Cell Carcinoma; PDT treatment; photodynamic therapy; Jet injection; Memorial Sloan Kettering Cancer Center; 20-270
MeSH Terms: conditions — Carcinoma, Basal Cell; Neoplasms, Basal Cell | interventions — Lighting; Infectious Disease Incubation Period

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tumor Excision, No Illumination (Experimental): The first four patients will not receive illumination but have their tumors excised after jet-injection (AirGent2.0) of ALA (Levulan Kerastick), and 3h incubation; this will be done to assess biodistribution of ALA through fluorescence microscopy.
  Interventions: Drug: Jet injection of ALA; Procedure: Surgical excision; Other: Incubation
- PDT treatment with jet-injections (Experimental): Patient 5-16 will receive PDT treatment with jet-injections of ALA followed by 3h incubation under occlusion and thereafter illumination with red light (total dose 75 J/cm2). In patient 5-16, the PDT treatment will be repeated after 2 weeks.
  Interventions: Drug: Jet injection of ALA; Procedure: Surgical excision; Procedure: Illumination; Other: Incubation

INTERVENTIONS:
Drug: Jet injection of ALA — The Basal Cell Carcinoma/BCC tumor and a 5 mm margin will be injected with a grid of 80 microliters of 20% ALA at 5-8.5 mm between each injection (30-50% overlap).
Procedure: Surgical excision — In the first 4 patients, the tumor will be excised according to national guidelines after 3h incubation (+/- 30 min is accepted).
Procedure: Illumination — For patients 5-16,after 3h incubation (+/- 30 min), the tumor will be illuminated with red light corresponding to a dose of 75 J/cm2 570- 670 nm or equivalent dose of narrowband red light. The intervention will be repeated at after 14 days in patient 5-16. If the wound is not healed at two weeks, the treatment may be postponed to allow healing (patient 5-16).
  Arms: PDT treatment with jet-injections
Other: Incubation — After injection of ALA, the tumor will be occluded with a light proof dressing and incubated for 3h (+/- 30 min).

SUMMARY:
The purpose of this study is to find out whether injecting ALA into the skin with a jet-injection device and activating the drug with light is a safe treatment that causes few or mild side effects in people with basal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria are eligible to participate in this study

* Histologically-verified, previously untreated low-risk mixed superficial and nodular BCC(s) or nodular BCC(s) < 1 cm in diameter on scalp, extremities, or trunk.
* ≥ 18 years of age
* Owner of a smartphone (Android or iPhone). Patients without a working smartphone will not be considered eligible for this study.
* Being able to download application on their phone
* Being able to take pictures of their treated BCC(s) (with or without assistance)
* Female subjects of childbearing potential must be confirmed not pregnant by a negative urine pregnancy test prior to trial treatment. (Female subjects are considered of childbearing potential unless they have been hysterectomized or have undergone tubal ligation or have been post-menopausal for at least one year prior to the first visit)
* Legally competent, able to give verbal and written informed consent
* Subject in good general health and willing to participate comply with protocol requirements.
* Superficial and nodular BCC(s)

Exclusion Criteria:

Subjects meeting any one of the following criteria are not eligible to participate in this study

* High-risk BCC(s) (H area, >1 cm in M area, or >2 cm in L area)
* BCC(s) subtype morpheaform
* Diagnosed with gorlin syndrome
* Receiving immunosuppressive medication
* Subjects with a known allergy to ALA
* Individuals with other interfering skin diseases in the area of treatment
* Subjects with a tattoo in the treatment area which may interfere with or confound the evaluation of the study
* Subjects with a history of keloids which is deemed clinically relevant in the opinion of the investigator
* Lactating or pregnant women
* Patient who are taking prescription pain medications or can not stop OTC pain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of local skin responses on Day 0 | Day 1
  Clinical evaluation of local skin responses on a 0-4 point scale will be performed at Day 0 (PDT treatment #1)
Clinical evaluation of local skin responses on Day 3 | Day 3
  Clinical evaluation of local skin responses on a 0-4 point scale will be performed at Day 3
Clinical evaluation of local skin responses on Day 14 | Day 14
  Clinical evaluation of local skin responses on a 0-4 point scale will be performed at Day 14 (PDT treatment #2)
Clinical evaluation of local skin responses on Day 17 | Day 17
  Clinical evaluation of local skin responses on a 0-4 point scale will be performed at Day 17
Clinical evaluation of local skin responses 3 months post treatment | 3 months after treatment
  Clinical evaluation of local skin responses on a 0-4 point scale will be performed 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Rossi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org